CLINICAL TRIAL: NCT01922583
Title: A Multi-center Phase II Study of AUY922 in Patients With Stage IV Non-small Cell Lung Cancer (NSCLC) With Driver Molecular Alterations Other Than Sensitive EGFR Mutation, Who Have Progressed After One Line of Systemic Therapy
Brief Title: AUY922 in Patient With Stage IV NSCLC
Acronym: NSCLC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAUY922ATW02T(201302063MIPD); 1020009413 (Other: Taiwan Food and Drug Administration (TFDA))
Record Dates: First submitted 2013-08-02; First posted 2013-08-14 (Estimated); Last update posted 2018-07-18 (Actual); Status verified 2017-02

CONDITIONS: Non-small Cell Lung Cancer (NSCLC)
Keywords: NSCLC, EGFR mutation
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — 5-(2,4-dihydroxy-5-isopropylphenyl)-4-(4-morpholin-4-ylmethylphenyl)isoxazole-3-carboxylic acid ethylamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vial (Experimental): AUY922 will be administered via IV over 1 hour once weekly in a 21 day cycle until disease progression
  Interventions: Drug: AUY922

INTERVENTIONS:
Drug: AUY922 — AUY922 will be administered via IV over 1 hour once weekly in a 21 day cycle until disease progression

SUMMARY:
This is an open-label, single-arm, multicenter phase II trial in patients with stage IV EGFR T790M, EGFR exon 20 and other uncommon, HER2, or BRAF-mutated; ALK, ROS1, or RET-rearranged NSCLC.

DETAILED DESCRIPTION:
Study Design:

This is an open-label, single-arm, multicenter phase II trial in patients with stage IV EGFR T790M, EGFR exon 20 and other uncommon, HER2, or BRAF-mutated; ALK, ROS1, or RET-rearranged NSCLC (n = 9 x 7)

Objectives:

Primary objective(s):

To define the objective response rate by RECIST 1.1 of AUY922 in patients with stage IV EGFR T790M, EGFR exon 20 and other uncommon, HER2, or BRAF-mutated; ALK, ROS1, or RET-rearranged NSCLC

Secondary objective(s):

(1) To define the disease control rate (complete response + partial response + stable disease >=24 weeks) of AUY922 in patients with stage IV EGFR T790M, EGFR exon 20 and other uncommon, HER2, or BRAF-mutated; ALK, ROS1, or RET-rearranged NSCLC. (2) To determine the progression-free survival of AUY922 in patients with stage IV EGFR T790M, EGFR exon 20 and other uncommon, HER2, KRAS, or BRAF-mutated; ALK, ROS1, or RET-rearranged NSCLC. (3) To determine the overall survival of AUY922 in patients with stage IV EGFR T790M, EGFR exon 20 and other uncommon, HER2, KRAS, or BRAF-mutated; ALK, ROS1, or RET-rearranged NSCLC.

Exploratory Objective(s):

To study the pharmacodynamics of circulating tumor cells and plasma proteins.

Planned number of subjects: A total of 63 patients for the first stage of this study in 1 - 3 centers in Taiwan.

Patient population:

1. Stage IV (by AJCC 7th edition) NSCLC.
2. EGFR T790M mutation; EGFR exon 20 and other uncommon mutation; HER2 mutation; BRAF mutation; ALK translocation; ROS1 translocation; or RET translocation in tumor samples.
3. One line of prior systemic therapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically proven diagnosis of stage IV NSCLC (AJCC 7th) which had been treated with one systemic therapy.
* One of the molecular alterations as follows:

  * EGFR mutations in exon 20 T790M.
  * EGFR mutations in exon 20; in-frame duplication and/or insertion (e.g. A767_V769dupASV or H773_V774insH) or point mutations other than T790M; or other uncommon mutations.
  * HER2 mutation in exon 20; in-frame duplication and/or insertion (e.g. YVMA 776-779 ins).
  * BRAF mutation in exon 15; point mutation (e.g. V600E) or in exon 11; point mutation (e.g. G469A, D594G).
  * ALK translocation resulting in EML4-ALK, KIF5B-ALK, or TFG-ALK fusion as determined by an ALK break apart FISH assay and defined by an increase in the distance of 5' and 3' ALK probes (split 5'-3') or the loss of the 5' probe (single 3'). Positive ALK results from other methods such as immunohistochemistry (IHC) or reverse transcriptase polymerase chain reaction testing may also be acceptable.
  * ROS1 translocation resulting in CD74-ROS1 or SLC34A2-ROS1, etc.
  * RET translocation resulting in KIF5B-RET fusion, etc.
* Patients with brain metastases are eligible if treated and neurologically stable for at least 2 weeks and is not taking any steroid.
* Any prior chemotherapy, targeted therapy (monoclonal antibodies), or major surgeries must have had completed at least 4 weeks before initiation of study medication. Any prior targeted therapy (tyrosine kinase inhibitors), radiotherapy or minor surgeries must have had completed at least 2 weeks before initiation of study medication. Any acute toxicity must have recovered to <=grade 1 (except for alopecia).
* Patients must have measurable or evaluable disease as per RECIST version 1.1.
* 20 years of age or older
* ECOG performance status 0-2
* Adequate organ function as defined by the following criteria:

  * Bone marrow function
  * Hemoglobin >=8.0 g/dL
  * Absolute neutrophil count (ANC) >=1500/uL
  * Platelets >=100,000/uL
  * Hepatic function
  * Serum aspartate transaminase (AST) and serum alanine transaminase (ALT) <=3.0 x upper limit of normal (ULN) or AST and ALT <=5.0 x ULN if there is liver metastasis
  * Total serum bilirubin <=1.5 x ULN Renal function
  * Creatinine <= 1.5 x ULN or creatinine clearance >=45 mL/min
* Able to communicate well with the investigator, to understand and comply with the requirements of the study. Understand and sign the written informed consent.
* Patients must use effective methods of contraception during the study period and for at least 90 days following study completion (excluding surgically sterile male patients, surgically sterile or postmenopausal female patients).

Exclusion Criteria:

* Currently on other therapeutic clinical trials
* Prior treatment of HSP90 inhibitors
* Any of the following within 3 months before initiation of study medication

  * Myocardial infarction
  * Unstable angina
  * Coronary artery bypass graft
  * Congestive heart failure NYHA functional class III or IV
  * Cerebral vascular accident
  * Transient ischemic attack
  * Uncontrolled hypertension at screening
* Ongoing cardiac arrhythmias of NCI CTCAE grade >=2
* Active infection requiring antibiotics
* Pregnancy or breast feeding
* Prior malignancy within the past 5 years (excluding non-melanoma skin cancer, cervical carcinoma in situ, superficial bladder cancer, and early prostate cancer).
* Active hepatitis B or C; positive HIV test result.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Objective response rate | Patients will be followed up for 2 years(post disease progression)
  To define the by RECIST 1.1 of AUY922 in patients with stage IV EGFR T790M, EGFR exon 20 and other uncommon, HER2, or BRAF-mutated; ALK, ROS1, or RET-rearranged NSCLC

SECONDARY OUTCOMES:
Efficacy, progression-free survival (PFS) | Patients will be followed up for PFS and OS for 2 years.(post disease progression)
  Patients will be followed for progression-free survival (PFS) and overall survival (OS) which will be analyzed by using a Kaplan-Meier curve.
  Patients will be followed up for PFS and OS for 2 years.
overall survival (OS) | Patients will be followed up for OS for 2 years.(post disease progression)
  Patients will be followed for overall survival (OS)

CONTACTS AND LOCATIONS:
Overall Officials: Chih-Hsin Yang, MD, PhD, Principal Investigator — National Taiwan University Hospital
Locations (3):
- Taiwan (3):
  - National Cheng Kung University Hospital, Tainan
  - Department of Oncology, National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei